CLINICAL TRIAL: NCT01333943
Title: Saphenous (Adductor Canal) Nerve Block Versus Femoral Nerve Block for Total Knee Arthroplasty: A Novel Approach for Postoperative Analgesia
Brief Title: Saphenous Nerve Block Versus Femoral Nerve Block for Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012-031
Record Dates: First submitted 2011-04-08; First posted 2011-04-12 (Estimated); Results first posted 2017-12-18 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-04

CONDITIONS: Total Knee Arthroplasty
Keywords: Total Knee Replacement; Regional Anesthesia; Quadriceps; Muscle Strength; Muscle Strength Dynamometer; Quadriceps muscle strength after regional anesthesia for TKA
MeSH Terms: interventions — Nerve Block; Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental (Experimental): Saphenous (Adductor Canal) Nerve Block
  Interventions: Procedure: Study Group: Experimental
- Control (Active Comparator): Femoral Nerve Block
  Interventions: Procedure: Control Group

INTERVENTIONS:
Procedure: Study Group: Experimental — The study group will receive the saphenous nerve block, at the level of the adductor canal. The block will be under ultrasound guidance. The local anesthetic will be 15 ml of 0.5% bupivicaine. The study group will also receive a combined spinal epidural, with 2.5 ml of 0.5% bupivacaine as the spinal agent. Additional drugs include anti-emetics, specifically Ondansetron (4 mg).
  Other Names: Saphenous (Adductor Canal) Nerve Block
  Arms: Experimental
Procedure: Control Group — The control group will receive the femoral nerve block. The block will be under ultrasound guidance. The local anesthetic will be 30 ml of 0.25% bupivicaine. The control group will also receive a combined spinal epidural, with 2.5 ml of 0.5% bupivacaine as the spinal agent. Additional drugs include anti-emetics, specifically Ondansetron (4 mg).
  Other Names: Femoral Nerve Block
  Arms: Control

SUMMARY:
Currently, the regional anesthetic standard of care for total knee replacement surgery is combined spinal/epidural, with or without a femoral nerve block, or FNB. Lasting approximately 18 hours, the FNB works by numbing the femoral nerve (and its branches), which is the major nerve controlling the knee joint. The femoral nerve also provides movement and sensation. While this regional anesthetic technique offers significant postoperative pain relief, it is possible that it may cause muscle weakness and increase patients' recovery time. Hence there is a need for an alternative technique, one that may help minimize postoperative pain as effectively as the FNB, while not causing weakness of the quadriceps muscle.

The saphenous nerve, a branch of the femoral nerve, provides sensation to the knee. Thus it is hypothesized that by "blocking" or anesthetizing the saphenous nerve with local anesthetic closer to where it branches off, the area around and below the knee will feel numb. Yet unlike with the FNB, the quadriceps muscle itself will still be able to function.

Patients will be randomized to receive FNB or saphenous nerve block. Quadriceps strength will be tested using a dynamometer before surgery (baseline), 6-8 hours following anesthesia administration, and on postoperative days 1 and 2. It is hypothesized that patients who receive FNB will experience a 50% decrease in quadriceps strength compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

* All patients ages 18-90 undergoing primary unilateral total knee arthroplasty
* Planned use of neuraxial anesthesia
* Ability to follow study protocol
* American Society of Anesthesiology (ASA) Class 1-3

Exclusion Criteria:

* Contraindication to a spinal or epidural anesthetic
* Chronic opioid use (defined as daily or almost daily use of opioids for >3 months)
* Hypersensitivity and/or allergy to local anesthetics
* Intraoperative use of any volatile anesthetic
* Patients with a pre-existing neuropathy on the operative limb
* Contraindication to a femoral nerve block or saphenous nerve block
* Allergy to any of the study medications
* Non-English speaking patients

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2011-03; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David H. Kim, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- [Background] Maffiuletti NA. Assessment of hip and knee muscle function in orthopaedic practice and research. J Bone Joint Surg Am. 2010 Jan;92(1):220-9. doi: 10.2106/JBJS.I.00305. PMID 20048117
- [Background] Bohannon RW. Measuring knee extensor muscle strength. Am J Phys Med Rehabil. 2001 Jan;80(1):13-8. doi: 10.1097/00002060-200101000-00004. PMID 11138949
- [Background] Capdevila X, Barthelet Y, Biboulet P, Ryckwaert Y, Rubenovitch J, d'Athis F. Effects of perioperative analgesic technique on the surgical outcome and duration of rehabilitation after major knee surgery. Anesthesiology. 1999 Jul;91(1):8-15. doi: 10.1097/00000542-199907000-00006. PMID 10422923
- [Background] Singelyn FJ, Deyaert M, Joris D, Pendeville E, Gouverneur JM. Effects of intravenous patient-controlled analgesia with morphine, continuous epidural analgesia, and continuous three-in-one block on postoperative pain and knee rehabilitation after unilateral total knee arthroplasty. Anesth Analg. 1998 Jul;87(1):88-92. doi: 10.1097/00000539-199807000-00019. PMID 9661552
- [Background] Kandasami M, Kinninmonth AW, Sarungi M, Baines J, Scott NB. Femoral nerve block for total knee replacement - a word of caution. Knee. 2009 Mar;16(2):98-100. doi: 10.1016/j.knee.2008.10.007. Epub 2008 Nov 28. PMID 19046884
- [Background] Horn JL, Pitsch T, Salinas F, Benninger B. Anatomic basis to the ultrasound-guided approach for saphenous nerve blockade. Reg Anesth Pain Med. 2009 Sep-Oct;34(5):486-9. doi: 10.1097/AAP.0b013e3181ae11af. PMID 19920424
- [Background] Akkaya T, Ersan O, Ozkan D, Sahiner Y, Akin M, Gumus H, Ates Y. Saphenous nerve block is an effective regional technique for post-menisectomy pain. Knee Surg Sports Traumatol Arthrosc. 2008 Sep;16(9):855-8. doi: 10.1007/s00167-008-0572-4. Epub 2008 Jun 24. PMID 18574578
- See also: This is the link to the Hospital for Special Surgery home website. — http://www.hss.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental | Control
Started | 47 | 47
Completed | 46 | 47
Not Completed | 1 | 0
Not completed — Known neuropathy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental | Control | Total
Number analyzed (Participants) | 46 | 47 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.0 (9.4) | 67.6 (11.3) | 67.8 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 29 | 53
  Male | 22 | 18 | 40
Region of Enrollment [Number; unit: participants]
  United States | 46 | 47 | 93

OUTCOME MEASURES:

1. Primary Outcome: Quadriceps Muscle Strength
Description: Measurements were made by a handheld dynamometer while patients perform isometric exercises. Results are presented in kilogram-force (kgF) units. One kgF is equal to 9.80665 N.
Time Frame: 48 hours following administration of anesthesia.
Measure: Mean (Standard Deviation); unit: kilogram-force
Arm/Group | Experimental | Control
Number analyzed (Participants) | 46 | 47
kilogram-force | 7.3 (5.4) | 2.2 (3.8)

2. Secondary Outcome: Total Opioid Usage
Description: Opioid consumption data were collected and converted to oral morphine equivalents.
Time Frame: Postoperative day 4.
Population: One patient was excluded from analysis due to a condition. Data from the remaining 93 patients were analyzed.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Experimental | Control
Number analyzed (Participants) | 46 | 47
mg | 36.6 (17.9) | 35.8 (20.7)

3. Secondary Outcome: NRS Pain Scores at Rest
Description: Patients rated pain on a scale of 0-10, with 0 representing no pain and 10 representing worst pain.
Time Frame: Postoperative day 4.
Population: One patient was excluded at the time of analysis, and the remaining 93 patients were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental | Control
Number analyzed (Participants) | 46 | 47
units on a scale | 1.7 (1.9) | 0.9 (1.8)

4. Secondary Outcome: Patient Satisfaction With the Nerve Block.
Description: Patient satisfaction was measured on a 0-10 scale (0=not satisfied; 10=very satisfied).
Time Frame: 24 hours following administration of anesthesia.
Population: One patient was excluded from analysis, and the remaining 93 patients were included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental | Control
Number analyzed (Participants) | 46 | 47
units on a scale | 8.8 (1.9) | 9.1 (1.7)

5. Secondary Outcome: Incidence of Postoperative Complications.
Time Frame: Postoperative day 4.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 46 | 47
Participants | 0 | 0

6. Secondary Outcome: Total Length of Hospital Stay
Time Frame: Total length of hospital stay
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Experimental | Control
Number analyzed (Participants) | 46 | 47
days | 3.7 (0.8) | 3.6 (0.8)

ADVERSE EVENTS:
Time Frame: 4 days after surgery
Arm/Group | Experimental | Control
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/47
Other Adverse Events (participants affected / at risk) | 0/47 | 0/47

LIMITATIONS AND CAVEATS:
The duration of analgesia from the ACB block is unclear and was not measured. Also, a large follow-up study is needed to investigate whether ACB improves rehabilitation, incidence of falls, and/or length of hospital stay.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes